CLINICAL TRIAL: NCT02476812
Title: The Positive Piggy Bank - A Positive Activities Intervention for Improving Functional Status in Patients With Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Afton Hassett, Psy.D., Associate Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00100068
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Piggy Bank (Experimental): Patients randomized to this group will meet with a research assistant who provides an overview of the intervention, explains the rationale for this treatment, and then gives the patients the instructions, piggy bank, and currency slips. Participants in this group will receive instructions. At the end of the monitoring period, 30 days, they are to "close their account" by opening the piggy bank and reviewing all of the slips of paper.
  Study personnel will contact patients within 72 hours to answer questions. Participants will also be contacted at 30 days to let patients know that they should read all of their currency slips in one sitting. They are also told that the intervention part of the study is over and are asked they complete the follow up questionnaires. Then, study personnel will call again to let the participant know that the second set of questionnaires will be arriving by mail.
  Interventions: Behavioral: Positive Piggy Bank
- Waitlist Control (No Intervention): The control group will serve to show the relative benefits of the Positive Piggy Bank intervention. Those in the control group who meet study criteria will also receive regular care after their epidural steroid injection (e.g., physician visits, medication maintenance, standard patient education). These patients will follow the same questionnaire follow up procedures as listed above including phone calls. The phone call at 72 hours will be to simply thank them for their participation in the study. At the end of the study period, approximately three months, Wait List control patients will also be offered the Positive Piggy Bank intervention along with the supportive phone calls. Should they choose to try the Positive Piggy Bank intervention, they will be required to return to the center to pick up supplies and receive instruction. They will also complete study questionnaires by mail at 30 days to assess intra-individual change.

INTERVENTIONS:
Behavioral: Positive Piggy Bank — Already noted.
  Arms: Positive Piggy Bank

SUMMARY:
Investigators will conduct a randomized controlled trial of a 30-day positive activities intervention, Positive Piggy Bank, compared to a Wait-List control group (Figure 2). Prior to their scheduled appointment to undergo epidural steroid injection, all patients meeting study criteria will be contacted by research staff to be invited to participate in this study. Those interested will be asked to arrive 45 minutes before their regularly scheduled appointment. At that time they will learn more about the study and provide informed consent if they choose to participate. Participants will then complete the study questionnaires and be randomized 1:1 to the Positive Piggy Bank condition (n=100) or the Wait List control group (n = 100). All participants will receive the usual treatment provided at the Back & Pain Center at the University of Michigan, Department of Anesthesiology (e.g., maintenance of medication regimen, standard office visits). Post-intervention (Day 30) and 2 months after that (Day 90), participants will complete the same questionnaires by mail. The primary outcome will be improved functional status, while secondary outcomes will be symptomatic (i.e., pain, fatigue and sleep) and related to mood and well-being. After the study period, the patients in the Wait List control will be offered the Positive Piggy Bank intervention and will be asked to complete one more set of questionnaires at 30 days by mail.

ELIGIBILITY:
Inclusion Criteria: Primary diagnosis of back pain and schedule to undergo an epidural steroid injection. :

1. ages 18 to 80;
2. able to read/understand English and give consent;
3. willing and able to comply with all aspects of study procedures;
4. if on antidepressants, medications stable for ≥4 weeks prior to study;
5. no plan to initiate a new non-pharmacological pain intervention during the 30-day study period (e.g., back surgery, physical therapy, cognitive-behavioral therapy);
6. if on pain medications, medications stable for ≥4 weeks prior to study and no plans to switch medications during the 30-day study period.

   -

Exclusion Criteria: Participants may meet all criteria above, but will be excluded under the following additional conditions:

1. having a known psychotic disorder or the presence of another psychiatric condition (e.g., severe depression, suicidal ideation) or cognitive impairment (e.g., severe dyslexia, traumatic brain injury) limiting ability to give consent and/or participate fully in the study;
2. currently undergoing psychotherapeutic care at the Back & Pain Center;
3. other factors that at the discretion of the investigators would adversely affect study participation. We will not exclude participants who undergo unanticipated changes in treatment, but will handle these data as described later.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in functional status measured by Oswestry Disability Questionnaire | 2 months post intervention
  Change in functional status

CONTACTS AND LOCATIONS:
Locations (1):
- Back & Pain Center, University of Michigan, Ann Arbor, Michigan, United States